CLINICAL TRIAL: NCT04198649
Title: Effect of Azithromycin on Failure Proportion of Severe Periodontitis Non-surgical Treatment
Acronym: AZITHROPARO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: not enough patients
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6996
Record Dates: First submitted 2019-12-12; First posted 2019-12-13 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Severe Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azithromycin (Experimental): 62 patients Non-surgical periodontal treatment and two 250mg azithromycin tablets one time daily for 3 days
  Interventions: Drug: Non-surgical periodontal treatment and azithromycin treatment
- Placebo (Placebo Comparator): 62 patients Non-surgical periodontal treatment and two 250mg starch tablets one time daily for 3 days
  Interventions: Other: Non-surgical periodontal treatment and placebo treatment

INTERVENTIONS:
Drug: Non-surgical periodontal treatment and azithromycin treatment — Procedure: periodontal treatment: oral hygiene instruction, scaling and root planning Drug: two 250mg azithromycin tablets one time daily for 3 days after scaling and root planning sessions
  Arms: Azithromycin
Other: Non-surgical periodontal treatment and placebo treatment — Procedure: periodontal treatment: oral hygiene instruction, scaling and root planning Placebo: two 250mg starch tablets one time daily for 3 days after scaling and root planning sessions
  Arms: Placebo

SUMMARY:
Primary purpose: Evaluate the effect of azithromycin on failure proportion of severe chronic periodontitis non-surgical treatment; failure characterized by the persistence of at least one periodontal pocket> 5mm at 6 months

Secondary purpose:

* Evaluate the effect of azithromycin on the persistence of pathological periodontal pockets > 5mm during non-surgical treatment of severe chronic periodontitis at 3 months and 6 months
* Evaluate the effect of azithromycin on the changes of clinical signs, periopathogen levels, expression of macrolides resistance genes, and expression of antimicrobial peptides (PAMs) during treatment of severe chronic periodontitis at 3 months and 6 months
* Assess therapeutic observance and side effects of antibiotic treatment
* Assess at 3 and 6 months the potential interactions of local, bacterial (periopathogen and resistance gene) clinical factors, and host defense (PAMs) with the effect of azithromycin, on failure proportion of severe chronic periodontitis non-surgical treatment

ELIGIBILITY:
Inclusion Criteria:

* Patient with severe generalized chronic periodontitis (loss of attachment ≥ 5mm at > 30% sites) (AAP classification 1999) and periodontal pockets >5mm on at least 5% of sites
* presence of bleeding on probing (≥ 30%)
* male or female subject older than 35 Years
* patient with at least 15 teeth including at least 2 molars (excluding wisdom teeth)
* patient with social assurance
* voluntary patient who signed informed consent

Exclusion Criteria:

* Patient with contraindications to treatment with azithromycin or its excipient: absolute contraindications are the history of allergy to macrolides or one of the excipients used in this study, association with ergot derivatives Rye, Cisapride, colchicine, and severe hepatic deficiencies. Other contraindications are for patients at risk of cardiac arrhythmia (diagnosis of QT interval prolongation and/or concomitant treatments, electrolytic disorder (hypokalemia, hypomagnesemia, cardiac arrhythmia, heart failure), severe renal failure, and drug associations (Antivitamin K, statins)
* Patient with aggressive periodontitis (AAP classification 1999)
* Patient smoking more than 10 cigarettes/day
* Patient with endocarditis risk or requiring antibiotic prophylaxis
* Patient with antibiotic treatment within 6 months prior to periodontal examination
* Patient with anti-inflammatory treatment in the month preceding periodontal examination and/or anti-inflammatory treatment of more than 3 consecutive days in the 3 months preceding periodontal examination
* Patient following or having followed a drug treatment (cyclosporine and other anti-rejection drugs, antiepileptic, calcium inhibitor) influencing periodontal status
* Patient with pathologies influencing periodontal status and/or systemic or local inflammatory response, such as diabetes, infectious stomatitis or not, diseases inflammatory and autoimmune, immuno-depression
* Patient with prolonged oral hygiene disability (physical/psychic impossibility of brushing teeth)
* Patient with impaired oral condition (untreated cavities, non-dental teeth rehabilitated), dental infections whose management requires antibiotic treatment within 6 months
* Patient having specialized periodontal treatment, root planning, or a periodontal surgical treatment in the year prior to the examination
* Pregnant woman or breastfeeding
* Patient with repeated chronic infections (more than 3 times per year) requiring antibiotic treatment
* Patient who had oral antiseptic treatment in the previous month
* Patient included in another intervention research protocol or in periods of exclusion (participation in an observational study remains possible)
* Patient with high bleeding risk and/or INR > 4.
* Patient under guardianship and under protection of justice
* Patient unable to cooperate or understand the instructions related to the study and care

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with failure of treatment, failure defined by persistence of at least one residual periodontal pocket > 5mm | At 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France